CLINICAL TRIAL: NCT03323723
Title: Rinovum Subsidiary 2, LLC: Disposable Stress Urinary Incontinence Pessary Device Efficacy and Safety Study
Brief Title: Disposable Stress Urinary Incontinence Pessary Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rinovum Women's Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-00002
Record Dates: First submitted 2017-10-13; First posted 2017-10-27 (Actual); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Efficacy and Safety Study, Single Group, Open Study, Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RS-2 SUI Device (Other): Comparing use of device to non-treatment phase
  Interventions: Device: SUI Device

INTERVENTIONS:
Device: SUI Device — Pessary SUI device

SUMMARY:
This study is an interventional, single arm, multi-center study. It will be conducted at sites in the northeastern United States. The protocol will be approved by Chesapeake IRB or applicable local IRBs. The sample size will consist of approximately 50 participants. Participants will undergo an initial control period in which preweighed pads will be worn for 7 consecutive days for 12 hours. This will be followed by device usage for 14 consecutive days where participants will wear both device and preweighed pads simultaneously. for 12 hours.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of an over-the-counter (OTC) disposable stress urinary incontinence (SUI) pessary device. Specifically, this study will evaluate the effectiveness of the pessary device by assessing reduction in urine leakage in approximately 50 women with Stress Urinary Incontinence (SUI). Efficacy will be assessed by mean pad weight gain per hour, reduction of stress urinary incontinence events per day, and a quality of life questionnaire. The safety of the OTC SUI pessary device will be evaluated by assessing all adverse events, including the results of urinalysis, vaginal swab, and vaginal examination.

ELIGIBILITY:
Inclusion Criteria:

* • Provision of signed and dated informed consent form

  * Literacy must be in English (able to read and understand Informed Consent)
  * Stated willingness to comply with all study procedures and availability for the duration of the study
  * Female, aged >18
  * Be in generally good heath as determined by the Investigator
  * Have a physician diagnosis of SUI that occurred prior to or during the screening visit of this study
  * Have a > 3-month history of experiencing > 3 episodes of SUI per week
  * Be willing to use the investigational pessary device for the control of urinary incontinence
  * Have experience with wearing a tampon
  * The most recent Pap smear is normal within 36 months.

Exclusion Criteria:

* • Is pregnant, or planning to become pregnant during the study

  * Has been physician diagnosed with urge urinary incontinence or mixed urinary incontinence prior to or during the screening visit for this study
  * Is post-partum within 3 months
  * Has had an intrauterine device (IUD) placement of less than 6 months
  * Has self-reported difficulty emptying her bladder;
  * Has a history of Toxic Shock Syndrome (TSS) or symptoms consistent with TSS;
  * Has experienced difficulty inserting or wearing an intra-vaginal device, including a tampon;
  * Has had vaginal surgery, perineal surgery, uterine surgery, or abortion (spontaneous or induced) within the past 3 months;
  * Has any Screening laboratory value outside the laboratory reference range considered clinically significant by the Investigator which could impact the safety of the participant or the outcome of the study
  * Has an active urinary tract infection or vaginal infection requiring treatment
  * If for any reason, the Investigator decides that the participant should not participate in the study.
  * Class III Obesity (BMI> 40.0 kg/m2)
  * Advanced prolapse
  * Fit assessment is not successful during screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 73 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Felipe Duenas Garcia, MD, Principal Investigator — West Virginia University Medicine
Locations (3):
- United States (3):
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny Health Network/East Suburban OB/GYN, Monroeville, Pennsylvania
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duenas-Garcia OF, Shapiro RE, Gaccione P. Safety and Efficacy of a Disposable Vaginal Device for Stress Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2021 Jun 1;27(6):360-364. doi: 10.1097/SPV.0000000000000861. PMID 32453209

RESULTS

PARTICIPANT FLOW:
Groups:
- RS-2 SUI Device: All participants underwent a baseline phase, followed by a two week treatment phase wearing the RS-2 SUI pessary for 14 consecutive days, 12 hours per day. Treatment phase leakage was then compared to baseline leakage for each individual patient to evaluate change in leakage while wearing RS-2 device.
Period: Screening
Arm/Group | RS-2 SUI Device
Started | 73
Completed | 64
Not Completed | 9
Period: Baseline Phase
Arm/Group | RS-2 SUI Device
Started | 64
Completed | 60
Not Completed | 4
Period: Treatment Phase
Arm/Group | RS-2 SUI Device
Started | 60
Completed | 51
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Analysis conducted on mITT population.
Arm/Group | RS-2 SUI Device
Number analyzed (Participants) | 73
Age, Customized [Mean (Standard Deviation); unit: years] — Population: All analyses performed on mITT population.
  years
    Average Age: number analyzed (Participants) | 48
    Average Age | 53.4 (12.04)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, Female | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All analyses performed on mITT population.
  Participants
    number analyzed (Participants) | 48
    Hispanic or Latino | 5
    Not Hispanic or Latino | 43
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage Reduction of Mean Pad Weight Gain (g/hr) During Treatment Phase as Compared to Baseline Phase.
Description: Pad weight gain (PWG) was measured by weighing used pads returned by participants and subtracting the pre-weight of that pad to obtain the total weight of leakage. The total weight of leakage was then divided by the number of hours the pad was worn by the participant to calculate the PWG/hr. The average PWG/hr for baseline was calculated by averaging the PWG/hr for the entire 7 days of the baseline phase. The average treatment PWG/hr for treatment phase was calculated by averaging the PWG/hr of the last 7 days of treatment phase. The percent change from baseline to treatment phase was then calculated. The objective was to show that PWG/hr is reduced by >50% during treatment phase. Thus, the null hypothesis is that the mean weight gain reduction per hour is <=50%, and the alternative is that it is >50%, from the control period (no device) to the treatment period (women wearing the device).
Time Frame: 7 days of the baseline phase and 7 days of treatment phase
Population: mITT Population
Measure: Mean (98.33% Confidence Interval); unit: percent change
Arm/Group | RS-2 SUI Device
Number analyzed (Participants) | 48
percent change | -47.4 [-61.13 to -33.76]

2. Secondary Outcome: Change in Mean SUI Episodes During Treatment Phase as Compared to Baseline Phase
Description: Change in mean number of SUI episodes per day from the 7-day baseline period to the last 7 days of the 14-day device treatment period. Participants will record SUI episodes in the Study Diary during the baseline (7 days) and treatment (14 days) periods. Negative values are indicative of efficacious outcome. Each subject will have a change in the number of episodes per day from the control period to the treatment period. Specifically, the number of episodes will be recorded each day in the diary. For the control phase, there will be (at most) 7 days of data. The mean number of SUI episodes per day will be computed for each subject. The same measures will occur in the treatment period for the analysis period, the last 7 days.
Time Frame: 7 days of baseline period and last 7 days of treatment phase
Population: mITT population
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | RS-2 SUI Device
Number analyzed (Participants) | 48
number of episodes | -1.00 [-1.37 to -0.75]

3. Secondary Outcome: Change in Quality of Life From Before Treatment Phase to After Treatment Phase
Description: Change in Quality of Life as measured by the ICIQ-LUTSqol - The Quality of Life Questionnaire to be performed at baseline, before, and after treatment phase of the study is based on 20 questions referring to areas which may have been influenced or changed by accidental urine loss and/or prolapse. These questions are assigned a value of, 1 = 'Not at all,' 2= 'Slightly,' 3 = 'Moderately,' or 4 'A lot.' Each area is then assessed on a scale of 1-10 to see how much it bothers them. The Questionnaire is scored by taking the average score of items and then multiplying that value by 25 to put scores on a scale from 0 to 100. A lower score is considered less impact to quality of life and a higher score reflects more impact to quality of life. In the same manner, a reduction in scores at the end of the Treatment Phase from post-baseline/before Treatment Phase, reflects improved quality of life. A reduction in score of > 3.7 is considered the Minimum Clinically Important Difference (MCID).
Time Frame: Before Treatment Phase and After Treatment Phase is complete
Population: mITT population
Measure: Mean (95% Confidence Interval); unit: Change in QoL score
Arm/Group | RS-2 SUI Device
Number analyzed (Participants) | 48
Change in QoL score | -4.35 [-6.22 to -2.49]

4. Secondary Outcome: Adverse Events and Labs Evaluation to Determine Safety of the Device
Description: Evaluation and analysis of AEs to determine safety as recommended in FDA SUI Clinical Trial Guidance - The safety of the OTC SUI pessary device will be evaluated by assessing all adverse events, including the results of urinalysis, vaginal swab, and vaginal examination.
Time Frame: 21 days
Population: Safety population
Measure: Number; unit: events
Arm/Group | RS-2 SUI Device
Number analyzed (Participants) | 73
events
  Adverse Events | 40
  Abnormal Laboratory Findings | 3

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 21 days.
Arm/Group | RS-2 SUI Device
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 22/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RS-2 SUI Device (N=73)
General Disorders and Administration Site Conidtions - Other, Specify (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal and Urinary Disorders - Other, Specify (Asymptomatic Bacteruria) (Renal and urinary disorders) | 1 (1)
Renal and Urinary Disorders - Other, Specify (Nocturia) (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Genital Edema (Reproductive system and breast disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Uterine Pain (Reproductive system and breast disorders) | 4 (4)
Vaginal Discharge (Reproductive system and breast disorders) | 2 (2)
Vaginal Dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal Hemorrhage (Spotting) (Reproductive system and breast disorders) | 4 (4)
Vaginal Pain (Reproductive system and breast disorders) | 6 (14)
Pain of Skin (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research results and associated data will be considered confidential until the earlier of: (i) the first publication or presentation thereof data according to the terms of this agreement; (ii) one (1) year after conclusion, abandonment, or termination of the Research at all sites.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03323723/Prot_SAP_000.pdf